CLINICAL TRIAL: NCT02817061
Title: Effectiveness of Light for Enhancement of Cognition by Transcranial Repeated Application (ELECTRA): a Placebo-Controlled Study of Efficacy, Tolerability and Acceptability in Healthy Adult Volunteers
Brief Title: Effectiveness of Light for Enhancement of Cognition by Transcranial Repeated Application (ELECTRA)
Acronym: ELECTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Director, Wellman Center for Photomedicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016P001134
Record Dates: First submitted 2016-06-16; First posted 2016-06-29 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Disease Type and/or Category Not Applicable
Keywords: no keywords for disease type and/or category

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NIR brain stimulation (Experimental): An Omnilux device will be used to put NIR light on the head and forehead of the subject age 18-25 or 65-85. The device is a low risk device as determined by the IRB. Thirty (30) subjects will receive this light at 6 visits over 16 weeks.
  An automated interactive software self-test will be used at baseline and at three subsequent visits to quantify subject cognitive functions.
  Interventions: Device: Omnilux
- Sham (Sham Comparator): An Omnilux Device will be used at a safe wavelength not associated with photobiomodulation, putting sham light on the head and forehead of the subject age 18-25 or 65-85. The device is a low risk device as determined by the IRB. Thirty (30) subjects will receive this light at 6 visits over 16 weeks.
  An automated interactive software self-test will be used at baseline and at three subsequent visits to quantify subject cognitive functions.
  Interventions: Device: Omnilux

INTERVENTIONS:
Device: Omnilux — The Omnilux LED array sources can be changed to emit different wavelength.

SUMMARY:
Aim: Investigate whether transcranial photobiomodulation (tPBM) using near-infrared light exposure to the head, can improve frontal lobe executive function, working memory and overall mood in normal volunteer participants.

Hypothesis: The investigators predict that tPBM will increase cognitive functioning, as measured by Cambridge Cognition cognitive testing in study subjects.

DETAILED DESCRIPTION:
Photobiomodulation (PBM), also called low-level light therapy (LLLT), uses optical power densities less than 100 mW/cm², and usually in the red (600-700 nm) or near infrared (NIR) 780-1000 nm wavelength range. Different light sources (coherent lasers or non-coherent LEDs) used for PBM have been shown to produce beneficial cellular effects and to be responsible for preservation and recovery of tissue function in controlled trials in a wide range of disorders typified by stress injury or degeneration. During PBM, absorption of red or near-infrared photons by cytochrome c oxidase in the mitochondrial respiratory chain causes an increase in cellular respiration that continues for much longer than the light is present when delivered at appropriate fluence and exposure durations.

Primary cellular effects include increases in mitochondrial activity and ATP levels, production of low levels of reactive oxygen species, induction of transcription factors (including the pro- survival NF-kB), and inhibition of apoptosis.

Over the past decade several studies have reported that a single, transcranial PBM treatment at 810 nm delivered to the head had significant, beneficial effect when used to treat acute ischemic stroke in several different animal models and also in human clinical trials. A similar approach was used to treat acute traumatic brain injury (TBI) in mice and in humans. Pathological examination of the mouse brains demonstrated up- regulation of brain-derived neurotrophic factor (BDNF) and stimulated neurogenesis in the hippocampus and increased synaptogenesis in the cortex.

A clinical trial is currently in progress at MGH to treat persons with acute moderate TBI. Several studies have shown improvement of cognitive function in persons with chronic TBI. Studies have also been conducted in animal models and in persons with Alzheimer's disease, Parkinson's disease, depression and anxiety.

Only a very limited number of studies have so far been carried out to test NIR photobiomodulation in normal experimental rodents and in normal human volunteers.

In this study, an LED array light source will be used that has been cleared by the FDA for other human uses.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-25 or 65-85
* Women of child-bearing potential, must use a double-barrier method for birth control (e.g. condoms with spermicide) if sexually active during the study and for 30 days post treatment of any kind.
* Subject Informed Consent obtained in writing in compliance with local regulations prior to enrollment into this study.
* The subject (and caregiver, if applicable) is willing to participate in this study for at least 12 weeks.

Exclusion Criteria:

* Inability to speak or read English (necessary for cognitive testing software use).
* Pregnancy or lactation
* History of stroke or traumatic brain injury
* Substance dependence or abuse in the past 6 months
* Diagnosis with major psychiatric disease (Psychotic disorder or psychotic episode, bipolar affective disorder)
* Diagnosed with a neurodevelopmental condition (autism or ADHD)
* A traumatic event that resulted in PTSD
* Any unstable medical illness (defined as any medical illness which has not been well-controlled with standard-of-care medications)
* A significant skin condition (i.e., hemangioma, scleroderma, rash, open wound) or medical implant (e.g. metal plate, implantable shunt or valve) on the head.
* Inability to understand or participate in the consent and performance of the study.
* Those with Parkinson's Disease, End Stage Renal Disease, and/or End Stage Liver Disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
ERT: Emotional Recognition Task | 16 weeks
  The median latency from stimulus onset to the subject's response button touch (i.e. emotion chosen) for all problems during assessment blocks.
PAL: Paired Associates Learning | 16 weeks
  The number of times the subject chose the incorrect box for a stimulus on assessment problems, plus an adjustment for the estimated number of errors they would have made on any problems, attempts and recalls they did not reach
RTI: Reaction Time | 16 weeks
  The mean duration between the onset of the stimulus and the release of the button. Calculated for correct, assessed trials where the stimulus could appear in any one of five locations.
RVP: Rapid Visual Information Processing | 16 weeks
  A' (A prime) is the signal detection measure of sensitivity to the target, regardless of response tendency (the expected range is 0.00 to 1.00; bad to good). In essence, this metric is a measure of how good the subject is at detecting target sequences.
SST: Stop Signal Task | 16 weeks
  The estimate of the length of time between the go stimulus and the stop stimulus at which the subject is able to successfully inhibit their response on 50% of the trials.
SWM: Spatial Working Memory | 16 weeks
  Between errors are defined as times the subject revisits a box in which a token has previously been found. This is calculated for trials of four, six and eight tokens.

CONTACTS AND LOCATIONS:
Overall Officials: R. Rox Anderson, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will only be shared within the study staff member on the approved Institutional Review Board MGH protocol and to the sponsor, the AFOSR

REFERENCES:
- [Background] Chung H, Dai T, Sharma SK, Huang YY, Carroll JD, Hamblin MR. The nuts and bolts of low-level laser (light) therapy. Ann Biomed Eng. 2012 Feb;40(2):516-33. doi: 10.1007/s10439-011-0454-7. Epub 2011 Nov 2. PMID 22045511
- [Background] Lapchak PA. Taking a light approach to treating acute ischemic stroke patients: transcranial near-infrared laser therapy translational science. Ann Med. 2010 Dec;42(8):576-86. doi: 10.3109/07853890.2010.532811. Epub 2010 Nov 1. PMID 21039081
- [Background] Huang YY, Gupta A, Vecchio D, de Arce VJ, Huang SF, Xuan W, Hamblin MR. Transcranial low level laser (light) therapy for traumatic brain injury. J Biophotonics. 2012 Nov;5(11-12):827-37. doi: 10.1002/jbio.201200077. Epub 2012 Jul 17. PMID 22807422
- [Background] Naeser MA, Hamblin MR. Traumatic Brain Injury: A Major Medical Problem That Could Be Treated Using Transcranial, Red/Near-Infrared LED Photobiomodulation. Photomed Laser Surg. 2015 Sep;33(9):443-6. doi: 10.1089/pho.2015.3986. Epub 2015 Aug 17. No abstract available. PMID 26280257
- [Background] Xuan W, Vatansever F, Huang L, Hamblin MR. Transcranial low-level laser therapy enhances learning, memory, and neuroprogenitor cells after traumatic brain injury in mice. J Biomed Opt. 2014;19(10):108003. doi: 10.1117/1.JBO.19.10.108003. PMID 25292167
- [Background] Xuan W, Agrawal T, Huang L, Gupta GK, Hamblin MR. Low-level laser therapy for traumatic brain injury in mice increases brain derived neurotrophic factor (BDNF) and synaptogenesis. J Biophotonics. 2015 Jun;8(6):502-11. doi: 10.1002/jbio.201400069. Epub 2014 Sep 8. PMID 25196192
- [Background] Farfara D, Tuby H, Trudler D, Doron-Mandel E, Maltz L, Vassar RJ, Frenkel D, Oron U. Low-level laser therapy ameliorates disease progression in a mouse model of Alzheimer's disease. J Mol Neurosci. 2015 Feb;55(2):430-6. doi: 10.1007/s12031-014-0354-z. Epub 2014 Jul 4. PMID 24994540
- [Background] Johnstone DM, Moro C, Stone J, Benabid AL, Mitrofanis J. Turning On Lights to Stop Neurodegeneration: The Potential of Near Infrared Light Therapy in Alzheimer's and Parkinson's Disease. Front Neurosci. 2016 Jan 11;9:500. doi: 10.3389/fnins.2015.00500. eCollection 2015. PMID 26793049
- [Background] Schiffer F, Johnston AL, Ravichandran C, Polcari A, Teicher MH, Webb RH, Hamblin MR. Psychological benefits 2 and 4 weeks after a single treatment with near infrared light to the forehead: a pilot study of 10 patients with major depression and anxiety. Behav Brain Funct. 2009 Dec 8;5:46. doi: 10.1186/1744-9081-5-46. PMID 19995444
- [Background] Michalikova S, Ennaceur A, van Rensburg R, Chazot PL. Emotional responses and memory performance of middle-aged CD1 mice in a 3D maze: effects of low infrared light. Neurobiol Learn Mem. 2008 May;89(4):480-8. doi: 10.1016/j.nlm.2007.07.014. Epub 2007 Sep 12. PMID 17855128
- [Background] Blanco NJ, Maddox WT, Gonzalez-Lima F. Improving executive function using transcranial infrared laser stimulation. J Neuropsychol. 2017 Mar;11(1):14-25. doi: 10.1111/jnp.12074. Epub 2015 May 28. PMID 26017772